CLINICAL TRIAL: NCT02243475
Title: Probing the Role of Sodium Channels in Painful Neuropathies: Observational Study
Brief Title: Probing the Role of Sodium Channels in Painful Neuropathies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Maastricht University (Other); Yale University (Other); University of Manchester (Other); Deutsche Diabetes Gesellschaft (Other); Centre National de la Recherche Scientifique, France (Other); Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: PROPANE STUDY
Record Dates: First submitted 2014-09-12; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Painful Peripheral Neuropathy; Painless Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — identification of novel mutations in the genes encoding for Nav1.7, Nav1.8, Nav1.9, Nav1.6, and Nav1.3 sodium channels
Oversight: Data Monitoring Committee: No

SUMMARY:
Neuropathic pain is a frequent feature of peripheral neuropathy causing a significant impact on patients' quality of life and health care costs. Not all individuals with neuropathy develop pain and it is not possible to predict who is more or less susceptible among those with similar risk exposure. Current inability to identify high-risk individuals hinders development and application of therapies to counteract neuropathic pain and to address targeted prevention strategies. Recently, the investigators Consortium has identified novel pathogenic mutations in genes encoding for two sodium channels (Nav1.7 and Nav1.8) known to play a critical role in the generation and conduction of action potentials in nociceptors and their terminal axons. This study was undertaken in a carefully selected group of patients with painful neuropathy using a candidate gene approach and directly revealed targets for new therapeutic strategies. This discover widened the spectrum of sodium channel-related pain disorders including conditions more common in the general population than those known so far. PROPANE STUDY, starting from the hypothesis of a common origin of neuropathic pain in a cohort of patients with predominantly small fibre neuropathy, aims to develop this original idea in a larger and well characterized study population, to provide evidence for the reliable stratification of patients at high risk and potential new treatments tailored on patients' clinical features, in order to improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of sensory neuropathy, including pure small fibre neuropathy (SFN), based on established clinical, nerve conduction study (NCS) and skin biopsy findings (Tesfaye et al. Diab Care 2010) caused by

  1. type 1 or type 2 diabetes (World Health Organization criteria) with stable metabolic control for >6 months (haemoglobin A1C <9%); or
  2. idiopathic aetiology after ruling out all known causes of neuropathy including vitamin deficiencies, malignancies, toxic, drugs

Exclusion Criteria:

* any other cause of neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: homogeneous cohorts of patients (age >18 years) with painful and painless diabetic or idiopathic sensory neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with novel mutations in the genes encoding for Nav1.7, Nav1.8, Nav1.9, Nav1.6, and Nav1.3 sodium channels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Lauria, MD, Study Chair — FINCB

REFERENCES:
- [Derived] Ziegler D, Strom A, Bonhof GJ, Kannenberg JM, Heier M, Rathmann W, Peters A, Meisinger C, Roden M, Thorand B, Herder C. Deficits in systemic biomarkers of neuroinflammation and growth factors promoting nerve regeneration in patients with type 2 diabetes and polyneuropathy. BMJ Open Diabetes Res Care. 2019 Nov 27;7(1):e000752. doi: 10.1136/bmjdrc-2019-000752. eCollection 2019. PMID 31803481
- [Derived] Puttgen S, Bonhof GJ, Strom A, Mussig K, Szendroedi J, Roden M, Ziegler D. Augmented Corneal Nerve Fiber Branching in Painful Compared With Painless Diabetic Neuropathy. J Clin Endocrinol Metab. 2019 Dec 1;104(12):6220-6228. doi: 10.1210/jc.2019-01072. PMID 31390004